CLINICAL TRIAL: NCT05711225
Title: The Effect of Smoking Cessation Intervention in Pregnancy According to the Web-Based Transtheoretic Model on Postpartum Smoking Relapse
Brief Title: Transtheoretic Model, Postpartum Smoking Relapse, Smoking Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semra YILMAZ (Other)
Responsible Party: Sponsor-Investigator, Semra YILMAZ, Research Assistant, Adiyaman University
Organization: Adiyaman University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: SYILMAZ
Record Dates: First submitted 2022-12-12; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Postpartum Smoking Relapse
Keywords: Transtheoretical Model; Web-based smoking cessation intervention

STUDY DESIGN:
Intervention Model Description: The research was conducted as a pretest-posttest control group experimental model.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The behavior stage was determined by applying the "Stages of Change Scale" (SCS) form to the pregnant women in the experimental group. The pre-test data from the women in the experimental group were obtained through the website through the Participant Introduction Form,"Behavior Change Process Scale" (BCPS), "Self-Efficacy Scale/Encouraging Factors Scale" (SES/EFS) and "Decision Balance Scale" (DBS) before watching the videos. In addition, FNDT was applied to women who smoked during pregnancy. Post-test data from the women in the experimental group were collected by having them fill out the postpartum part of the Participant Identification Form at the 4th week postpartum after watching the animation videos, and FNDT, SCS, BCPS/EFS and DBS forms for those who still smoke, on the website.
  Interventions: Behavioral: smoking cessation intervention given according to the web-based transtheoretic model during pregnancy on postpartum smoking relapse.
- Control group (No Intervention): The behavior stage was determined by applying the "Stages of Change Scale" (SCS) form to the women participating in the control group. The pre-test data of the women participating in the control group were applied via the Participant Identification Form, FNDT, SCS, BCPS/EFS and DBS and the FNDT form to those who continued to smoke during pregnancy. Post-test data from women in the control group were collected with the postpartum part of the Participant Identification Form at 4 weeks postpartum, FNDT, SCS, BCPS/EFS and DBS for smokers.

INTERVENTIONS:
Behavioral: smoking cessation intervention given according to the web-based transtheoretic model during pregnancy on postpartum smoking relapse. — Smoking cessation videos prepared according to the Web-Based Transtheoretic model A module was created on the web, with 5 sections, prepared by the researcher according to the Web-Based Transtheoretic model, for quitting smoking or for pregnant women who quit smoking to maintain this behavior. The modules are prepared in the form of animated videos in which the researcher is educational. Each module is arranged for an average of 5-10 minutes. Theoretical information about the content has been added under each video.
  Arms: Experimental group

SUMMARY:
The postpartum period is an important opportunity to improve maternal and fetal health by preventing smoking relapse in women. To achieve this goal, digital platforms, which are the latest technological developments are used. However, studies using digital platforms on smoking cessation and postpartum smoking relapse in pregnant women are limited in this area. The research was carried out to determine the effect of smoking cessation intervention prepared in line with the transtheoretic model on the digital platform, on preventing smoking relapse in the postpartum period. As a result of the research, it is thought that nurses will guide their professional practices with an evidence-based up-to-date approach.

DETAILED DESCRIPTION:
Smoking during pregnancy is the most important cause of preventable complications. Smoking has many negative effects on fetal development and well-being as well as women's health. Pregnancy and childbirth can motivate women to quit smoking. However, it is stated that the rate of failure to quit smoking is higher in women than in men, and the period of resumption of smoking is shorter after an attempt to quit. In a large-scale study conducted in 54 low- and middle-income countries, it is stated that the prevalence of any tobacco use during pregnancy is 2.6%, with the highest prevalence being 15% in Turkey. The rates of smoking during pregnancy differ in studies conducted in our country. Due to the stigma and blame for smoking, many women report not smoking during pregnancy. This situation may prevent the exact number of pregnant women who smoke and prevent smoking cessation intervention and treatment. In our country, the rate of smoking during pregnancy was determined as 11.9% by Tarhan and Yılmaz, and as 13% by Dilcen et al. Smoking during pregnancy has numerous adverse effects on the mother and fetus. Intrauterine growth retardation, low birth weight, placenta previa and abruption, premature rupture of membranes, perinatal mortality during pregnancy; For newborns, the risk of developing asthma disease, infantile colic, obesity and sudden infant death are among the negative effects of maternal smoking. Factors affecting smoking during pregnancy were determined as planned pregnancy, number of pregnancies, gestational week, number of living children, frequency of receiving prenatal care, smoking status of the spouse and passive smoking.

It has been reported that women continue to smoke in the postpartum period despite quitting during pregnancy. In a meta-analysis study, it was shown that 43% of women who quit smoking during pregnancy started smoking again in the postpartum 6th month. It is stated that women continue to smoke after birth because they believe that they can no longer have a direct effect on their children. It has been reported that this situation may be related to smoking, postpartum fatigue, and stress related to child care. In addition, it has been shown that resumption of smoking after birth is associated with various factors such as young age, smoking status of people around, low income, and early cessation of breastfeeding. For this reason, it is stated that smoking in women is a complex phenomenon that can be affected by specific experiences related to social relations, pregnancy and birth, and this may cause an increase in postpartum relapse rates in women who quit smoking during pregnancy.

When interventions that support smoking cessation and prevention of relapse from pregnancy to postpartum are evaluated, it is stated that pregnancy is a trigger for smoking cessation and this period should be seen as an opportunity for smoking cessation interventions. Different intervention methods are used to quit smoking. Cessation interventions include informing, cognitive and behavioral treatments, hypnosis, acupuncture, and pharmacological treatments. There is insufficient evidence regarding the efficacy and safety of nicotine replacement, which is one of the pharmacological treatments used in smoking cessation during pregnancy. Instead, other interventions that are effective in quitting smoking during pregnancy; consultancy, feedback, financial incentives, telephone support programs, digital platforms and similar applications can be used. Digital interventions, including mobile health interventions, are considered an innovative way to provide evidence-based smoking cessation support to a hard-to-reach population. The use of digital platforms, including telephone, video, websites or mobile application technologies, can be used effectively to quit smoking during pregnancy. In their study, Derksen et al. found that social networks had a positive effect on the attitudes of pregnant women towards smoking cessation. Dascal et al., in their study to prevent postpartum smoking relapse, found that digital smoking cessation intervention had a positive effect on preventing postpartum smoking.

ELIGIBILITY:
Inclusion Criteria:

* Don't have a smartphone
* Having the ability to use the Internet
* 32nd gestational week and below
* Reporting smoking at least two cigarettes per day in the 3 months before conception

Exclusion criteria from the study:

• Not watching videos within the scope of web-based intervention.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Measure 1- The Fagerström Test for Nicotine Dependence | 15 months
  The Fagerström Test for Nicotine Dependence was developed to determine the level of addiction to cigarettes.The scores that can be obtained from the scale range from 0 to 10. As addiction to cigarette increases, the score obtained from the scale increases.
  it was determined that the mean score of the scale decreased and the level of addiction decreased in the intervention group.
Measure 2- Behavior Change Process Scale | 15 months
  It reveals what processes the individual has experienced in the stages of behavior change.The lowest score that can be obtained from the scale is 22, and the highest is 110. The higher the score obtained from the scale, the higher the chance of success in changing behavior. The higher the score obtained from the scale, the higher the chance of success in changing behavior.
  It was determined that women in the intervention group had a higher chance of success in changing their smoking behavior.
Measure 3-Self-Efficacy Scale/Encouraging Factors Scale | 15 months
  The Self-Efficacy Scale/Encouraging Factors Scale shows the confidence that individuals have in order not to return to the harmful behavior they have changed when faced with difficult situations. The lowest score that can be obtained from the scale is 8 and the highest 40. A high score on the self-efficacy scale reveals the success of not smoking and quitting smoking despite encouraging factors. A high score on the Encouraging Factors Scale indicates that the probability of returning to the harmful behavior is high. The Encouraging Factors Scale is used with an answer format that is the opposite of the Self-Efficacy Scale.
  Despite the fact that the women in the intervention group faced stimulant situations, not returning to smoking behavior again shows that the power to resist is high.
Measure 4-Decision Balance Scale | 15 months
  The decision balance scale reveals the positive and negative perceptions of behavior change. The scale consists of two sub-dimensions that reveal the perception of the positive and negative aspects of smoking. The lowest score that can be obtained for the two sub-dimensions of the scale is 12, and the highest score is 60. A high score on the benefit (positive) sub-dimension indicates his indecision about changing behavior, while a high score on the harm (negative) sub-dimension indicates that has a higher chance of making and continuing a decision on behavior change.
  It was determined that women in the intervention group were more determined to change their smoking behavior and were more likely to maintain this determination.

CONTACTS AND LOCATIONS:
Overall Officials: SEMRA YILMAZ, Principal Investigator — Research Assistant
Locations (1):
- Semra YILMAZ, Merkez, Adıyaman Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loukopoulou AN, Vardavas CI, Farmakides G, Rossolymos C, Chrelias C, Tzatzarakis MN, Tsatsakis A, Lymberi M, Connolly GN, Behrakis PK. Design and study protocol of the maternal smoking cessation during pregnancy study, (M-SCOPE). BMC Public Health. 2011 Dec 6;11:903. doi: 10.1186/1471-2458-11-903. PMID 22145828
- [Background] Lanting CI, van Wouwe JP, van den Burg I, Segaar D, van der Pal-de Bruin KM. [Smoking during pregnancy: trends between 2001 and 2010]. Ned Tijdschr Geneeskd. 2012;156(46):A5092. Dutch. PMID 23151329
- [Background] Lange S, Probst C, Rehm J, Popova S. National, regional, and global prevalence of smoking during pregnancy in the general population: a systematic review and meta-analysis. Lancet Glob Health. 2018 Jul;6(7):e769-e776. doi: 10.1016/S2214-109X(18)30223-7. Epub 2018 May 31. PMID 29859815
- [Background] Scheffers-van Schayck T, Tuithof M, Otten R, Engels R, Kleinjan M. Smoking Behavior of Women Before, During, and after Pregnancy: Indicators of Smoking, Quitting, and Relapse. Eur Addict Res. 2019;25(3):132-144. doi: 10.1159/000498988. Epub 2019 Mar 27. PMID 30917383
- [Background] Caleyachetty R, Thomas GN, Toulis KA, Mohammed N, Gokhale KM, Balachandran K, Nirantharakumar K. Metabolically Healthy Obese and Incident Cardiovascular Disease Events Among 3.5 Million Men and Women. J Am Coll Cardiol. 2017 Sep 19;70(12):1429-1437. doi: 10.1016/j.jacc.2017.07.763. PMID 28911506
- [Background] Kahyaoğlu S, Özel Ş, Üstün YE, Erdöl C. Gebelik ve Sigara Bırakma. Jinekoloji-Obstetrik ve Neonatoloji Tıp Derg 2018, 15: 1.
- [Background] Tarhan P, Yılmaz T. Gebelikte sigara kullanımı ve etkileyen faktörler. Sağlık Bilimleri ve Meslekleri Derg 2016, 3(3): 140-7.
- [Background] Dilcen HY, Öztürk A, Yıldız MN. Gebelikte Sigara Kullanımının Algılanan Sosyal Destek, Benlik Saygısı ve Psikolojik Sağlamlık ile İlişkisi. Bağımlılık Derg 2021, 22(2): 161-70.
- [Background] Chamberlain C, O'Mara-Eves A, Porter J, Coleman T, Perlen SM, Thomas J, McKenzie JE. Psychosocial interventions for supporting women to stop smoking in pregnancy. Cochrane Database Syst Rev. 2017 Feb 14;2(2):CD001055. doi: 10.1002/14651858.CD001055.pub5. PMID 28196405
- [Background] Harmer C, Memon A. Factors associated with smoking relapse in the postpartum period: an analysis of the child health surveillance system data in Southeast England. Nicotine Tob Res. 2013 May;15(5):904-9. doi: 10.1093/ntr/nts221. Epub 2012 Oct 8. PMID 23045522
- [Background] Jones M, Lewis S, Parrott S, Wormall S, Coleman T. Re-starting smoking in the postpartum period after receiving a smoking cessation intervention: a systematic review. Addiction. 2016 Jun;111(6):981-90. doi: 10.1111/add.13309. Epub 2016 Mar 16. PMID 26990248
- [Background] Diamanti A, Papadakis S, Schoretsaniti S, Rovina N, Vivilaki V, Gratziou C, Katsaounou PA. Smoking cessation in pregnancy: An update for maternity care practitioners. Tob Induc Dis. 2019 Aug 2;17:57. doi: 10.18332/tid/109906. eCollection 2019. PMID 31582946
- [Background] Marufu TC, Ahankari A, Coleman T, Lewis S. Maternal smoking and the risk of still birth: systematic review and meta-analysis. BMC Public Health. 2015 Mar 13;15:239. doi: 10.1186/s12889-015-1552-5. PMID 25885887
- [Background] Notley C, Gentry S, Livingstone-Banks J, Bauld L, Perera R, Hartmann-Boyce J. Incentives for smoking cessation. Cochrane Database Syst Rev. 2019 Jul 17;7(7):CD004307. doi: 10.1002/14651858.CD004307.pub6. PMID 31313293
- [Background] Stead LF, Koilpillai P, Fanshawe TR, Lancaster T. Combined pharmacotherapy and behavioural interventions for smoking cessation. Cochrane Database Syst Rev. 2016 Mar 24;3(3):CD008286. doi: 10.1002/14651858.CD008286.pub3. PMID 27009521
- [Background] Herbec A, Beard E, Brown J, Gardner B, Tombor I, West R. The needs and preferences of pregnant smokers regarding tailored Internet-based smoking cessation interventions: a qualitative interview study. BMC Public Health. 2014 Oct 14;14:1070. doi: 10.1186/1471-2458-14-1070. PMID 25312556
- [Background] Tombor I, Neale J, Shahab L, Ruiz M, West R. Healthcare providers' views on digital smoking cessation interventions for pregnant women. J Smoking Cessat 2015, 10(2): 116-23.
- [Background] Derksen ME, Kunst AE, Murugesu L, Jaspers MWM, Fransen MP. Smoking cessation among disadvantaged young women during and after pregnancy: Exploring the role of social networks. Midwifery. 2021 Jul;98:102985. doi: 10.1016/j.midw.2021.102985. Epub 2021 Mar 11. PMID 33761432
- [Background] Dascal M, Rusu A, Onisor A, Blaga O, Miller M, Meghea C. An mHealth intervention to prevent postnatal smoking relapse: The RESPREMO study protocol. Tob Prev Cessat. 2020 Apr 14;6:24. doi: 10.18332/tpc/118724. eCollection 2020. PMID 32548361